CLINICAL TRIAL: NCT00101101
Title: A Phase II Trial Using a Universal GM-CSF-Producing and CD40L-Expressing Bystander Cell Line (GM.CD40L) in the Formulation of Autologous Tumor Cell-Based Vaccines for Patients With Mantle Cell Lymphoma
Brief Title: Universal Granulocyte Macrophage-colony Stimulating Factor (GM-CSF)-Producing and GM.CD40L for Autologous Tumor Vaccine in Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Lymphoma Research Foundation (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13840; 0406-654 (Other: OBA)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Lymphoma
Keywords: recurrent mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Dexamethasone; Calcium Dobesilate; Interleukin-2; Cytokines; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine and Conventional Therapy (Experimental): Patients were treated with 3-6 cycles of chemotherapy +/- rituximab, with type and duration at the discretion of the individual clinician.
  Chemotherapy: 6 courses of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) OR 3 courses of hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone alternating with high-dose methotrexate and cytarabine (hyper-CVAD) for patients who have relapsed after CHOP.
  Patients who achieve a partial or complete response after completion of chemotherapy proceed to autologous tumor cell-based vaccine therapy.
  Patients who have stable or responding disease at 12 months receive 4 additional courses of booster vaccine and low-dose IL-2.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Dexamethasone; Biological: Autologous Tumor Cell-Based Vaccine; Drug: IL-2

INTERVENTIONS:
Drug: Cyclophosphamide — Participants receive conventional chemotherapy comprising 6 courses of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) OR 3 courses of hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone alternating with high-dose methotrexate and cytarabine (hyper-CVAD) for patients who have relapsed after CHOP.
  Other Names: Cytoxan
Drug: Doxorubicin — Participants receive conventional chemotherapy comprising 6 courses of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) OR 3 courses of hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone alternating with high-dose methotrexate and cytarabine (hyper-CVAD) for patients who have relapsed after CHOP.
  Other Names: adriamycin; Rubex
Drug: Vincristine — Participants receive conventional chemotherapy comprising 6 courses of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) OR 3 courses of hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone alternating with high-dose methotrexate and cytarabine (hyper-CVAD) for patients who have relapsed after CHOP.
  Other Names: Oncovin; leurocristine; VCR
Drug: Prednisone — Participants receive conventional chemotherapy comprising 6 courses of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) OR 3 courses of hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone alternating with high-dose methotrexate and cytarabine (hyper-CVAD) for patients who have relapsed after CHOP.
  Other Names: Deltasone; Liquid Pred; Meticorten; Orasone
Drug: Dexamethasone — Participants receive conventional chemotherapy comprising 6 courses of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) OR 3 courses of hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone alternating with high-dose methotrexate and cytarabine (hyper-CVAD) for patients who have relapsed after CHOP.
  Other Names: Decadron; Dexasone; Diodex; Hexadrol
Biological: Autologous Tumor Cell-Based Vaccine — Participants receive vaccine comprising autologous tumor cells and GM.CD40L intradermally on day 1 and low-dose interleukin-2 (IL-2) subcutaneously twice daily on days 1-14. Treatment repeats every 28 days for 4 courses. Patients who have stable or responding disease at 12 months receive 4 additional courses of booster vaccine and low-dose IL-2 as above.
Drug: IL-2 — Participants receive vaccine comprising autologous tumor cells and GM.CD40L intradermally on day 1 and low-dose interleukin-2 (IL-2) subcutaneously twice daily on days 1-14. Treatment repeats every 28 days for 4 courses. Patients who have stable or responding disease at 12 months receive 4 additional courses of booster vaccine and low-dose IL-2 as above.
  Other Names: interleukin-2; cytokine; aldesleukin

SUMMARY:
RATIONALE: Vaccines made from gene-modified cells and a person's cancer cells may make the body build an effective immune response to kill cancer cells. Interleukin-2 (IL-2) may stimulate the white blood cells to kill cancer cells. Giving booster vaccinations may make a stronger immune response and prevent or delay the recurrence of cancer. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Giving vaccine therapy together with IL-2 after combination chemotherapy may be a more effective treatment for mantle cell lymphoma.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with IL-2 after combination chemotherapy works in treating patients with relapsed or de novo stage II, stage III, or stage IV mantle cell lymphoma.

DETAILED DESCRIPTION:
Patients were treated with 3-6 cycles of chemotherapy +/- rituximab, with type and duration at the discretion of the individual clinician. Evaluation for response was performed 1 month after completing chemotherapy, and included computed tomography (CT) scan, bone marrow biopsy, endoscopy, and colonoscopy. Minimal residual disease (MRD) was assessed qualitatively on bone marrow specimens using polymerase chain reaction (PCR) with standardized primers for evaluation for B-cell receptor gene rearrangement. Responses were defined according to revised Cheson criteria. Patients with successful lymph node harvest who had obtained complete or partial response could proceed to bystander vaccination.

The GM.CD40L bystander vaccine administered intradermally into the bilateral axillary and inguinal nodal basins via eight separate injections (0.125 ml / injection). Low dose IL-2 (0.5 x 10^6 units) was given subcutaneously twice daily for 14 days following vaccination. Patients were restaged with CT and/or CT/PET and bone marrow biopsy every 6 months, beginning from the last date of chemotherapy. Follow-up bone marrow biopsy evaluation included an assessment for MRD as described above. Patients without disease progression or toxicity attributable to the vaccine were eligible for 4 monthly booster vaccines at 12 months and 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mantle cell lymphoma

  * Stage II, III, or IV disease
  * Relapsed or de novo disease
* No symptomatic brain metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy

* Not specified

Hematopoietic

* White blood count (WBC) > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hematocrit > 25%
* Hemoglobin > 8 g/dL

Hepatic

* Bilirubin < 2.0 mg/dL

Renal

* Creatinine < 2.0 mg/dL OR
* Creatinine clearance > 60 mL/min

Immunologic

* No serious ongoing infection
* No known HIV infection
* No other pre-existing immunodeficiency condition

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 1 month before, during, and for 3 months after study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent immunotherapy

Chemotherapy

* More than 4 weeks since prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* More than 4 weeks since prior steroids
* No concurrent corticosteroids except as replacement doses in patients who are hypoadrenal

Radiotherapy

* More than 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No other concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Dessureault, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty three patients with stage II-IV histologically confirmed mantle cell lymphoma (MCL) in need of systemic chemotherapy were enrolled at the H. Lee Moffitt Cancer Center between February 2004 and July 2008.
Period: Overall Study
Arm/Group | Vaccine and Conventional Therapy
Started | 43
Completed | 23 (Participants who received at least one vaccine injection.)
Not Completed | 20
Not completed — never received vaccine | 20

BASELINE CHARACTERISTICS:
Population: All participants who started the study.
Arm/Group | Vaccine and Conventional Therapy
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 25
Age, Continuous [Median (Full Range); unit: participants] | 65 [47 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Rate of Immunological Response to Vaccination
Description: Immunological response to vaccination, as measured by in vitro testing of peripheral blood mononuclear cells (PBMCs) for interferon gamma secretion, delayed type hypersensitivity reaction (DTH) in response to irradiated autologous tumor cells, and lymphocyte accumulation at DTH and vaccine injection sites.
  DTH Skin Testing was performed within 2 weeks prior to first vaccine, and again after fourth vaccine was administered. Aliquots containing 10^6 irradiated autologous tumor cells were re-suspended in 0.2 mL of Plasma-Lyte A and injected intradermally in the forearm and marked. 48 hours later, injection site was inspected for induration and erythema.
  3mm punch biopsy of DTH injection site and vaccine site was obtained 48 hours after administration of irradiated tumor cells before and after the vaccine series. Vaccine site biopsy was obtained 2-5 days after the second vaccine had been given. Granulocytic and lymphocytic accumulation at these sites was graded by a pathologist.
Time Frame: 4 months per participant
Population: Participants who received at least one vaccine injection.
Measure: Number; unit: participants
Arm/Group | Vaccine and Conventional Therapy
Number analyzed (Participants) | 23
participants
  Clinical DTH | 0
  Increase in Interferon Gamma Secretion | 15

2. Secondary Outcome: Occurrence of Related Serious Adverse Events (SAEs)
Description: Patients were monitored for toxicity every 4 weeks in clinic throughout the 4-month vaccination phase. This included clinical and laboratory evaluation (CBC, blood urea nitrogen (BUN), creatinine, electrolytes, liver function test (LFT), and serum LDH). Toxicity was defined according to the NCI Common Terminology Criteria for Adverse Events (CTCAE-3) Version 3.0 (www.ctep.cancer.gov). Grade 3 or higher SAEs attributed to vaccination: Toxicity was assessed in the 23 patients who received at least one vaccine injection.
Time Frame: 4 months per participant
Population: Participants who received at least one vaccine injection.
Measure: Number; unit: participants
Arm/Group | Vaccine and Conventional Therapy
Number analyzed (Participants) | 23
participants | 0

3. Secondary Outcome: Median Event Free Survival (EFS)
Description: Vaccine Response - EFS among participants who received vaccination. Event free survival (EFS) was calculated from date of enrollment until progression or death from any cause. Progressive disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 18 months
Population: Participants who received at least one vaccine injection.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vaccine and Conventional Therapy
Number analyzed (Participants) | 23
months | 9 [5 to 18]

ADVERSE EVENTS:
Time Frame: Patients were monitored for toxicity every 4 weeks in clinic throughout the 4-month vaccination phase.
Arm/Group | Vaccine and Conventional Therapy
Serious Adverse Events (participants affected / at risk) | 2/43
Other Adverse Events (participants affected / at risk) | 11/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine and Conventional Therapy (N=43)
Leukocyte (Blood and lymphatic system disorders) | 1 (2)
Granulocyte (Blood and lymphatic system disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine and Conventional Therapy (N=43)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 11 (25)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 (10)
Fever (in the absence of neutropenia) (General disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 6 (6)
Platelets (Blood and lymphatic system disorders) | 3 (3)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (2)
Pain - Joint (General disorders) | 4 (4)
Pain - Head/headache (General disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
With a median follow-up of 67 months, the median overall survival (OS) has not yet been reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes